CLINICAL TRIAL: NCT00411268
Title: Safety, Efficacy and Impact on Quality of Life of Long-Term Administration of Dilaudid CR (Hydromorphone HCI) in Patients With Chronic Low Back Pain
Brief Title: Safety, Effectiveness, and Impact on Quality of Life on Long-Term Administration of OROS Hydromorphone Slow-Release in Patients With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013258
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2010-04-27 (Estimated); Status verified 2010-04

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; OROS hydromorphone slow release tablet; Quality of Life
MeSH Terms: conditions — Low Back Pain

INTERVENTIONS:
Drug: OROS hydromorphone HCI SR (slow release)

SUMMARY:
The purpose of this open-label, extension study is to characterize the safety, effectiveness, and impact on quality of life measures of long-term repeated dosing of OROS hydromorphone slow release (8, 16, 32 and 64 mg tablets) in patients with chronic low back pain.

DETAILED DESCRIPTION:
This open label, extension study characterized the safety, effectiveness, and impact on quality of life of OROS hydromorphone slow release with long-term repeated dosing among patients with chronic low back pain, who previously completed short-term Study DO-127 with OROS hydromorphone slow release. Up to 150 patients were to be enrolled and evaluated. Patients were enrolled in this study immediately following Study DO-127. Patients continued their therapy with OROS hydromorphone slow release at the stable dose previously identified in the short-term study. The patient's initial prescribed dose of OROS hydromorphone slow release in Study DO-127X was the same as the last dose of OROS hydromorphone slow release in Study DO-127. Patients returned monthly for evaluations during this extension interval. Adjustments to dose were performed as needed, at the Investigator's discretion. The duration of this study was six months. Safety assessments included vital signs and physical examination at start, during and end of study. 8, 16, 32 and 64 mg tablets of OROS hydromorphone (dose will be at Investigators' discretion) slow release tablets were taken orally daily for the duration of the six month study

ELIGIBILITY:
Inclusion Criteria:

* Patients who have chronic low back pain who have successfully completed short-term Study DO-127 with OROS hydromorphone slow release
* Patients who require at least 8 mg of hydromorphone HCI (slow release) every 24 hours for the management of chronic low back pain
* Patients whose opioid requirements have been stable as demonstrated in short-term Study DO-127 with OROS hydromorphone slow release

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid agonists)
* Patients who are pregnant or breast-feeding
* Patients with any gastrointestinal disorder, including pre-existing severe GI narrowing (pathologic or iatrogenic) that may affect the absorption or transit of orally administered drugs
* Patients with significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, disorders of cognition, any clinically significant impaired renal or hepatic function, Addison's disease, hypothyroidism, prostatic hypertrophy, or urethral stricture
* Patients who may be at risk for serious decreases in blood pressure upon taking an opioid analgesic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Study Completion 2001-06 (Actual)

PRIMARY OUTCOMES:
The daily pain relief rating obtained during the study.(six months)

SECONDARY OUTCOMES:
Differences from first visit to each subsequent visit in Brief Pain Inventory (BPI) ratings, sleep scores and quality of life questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA